CLINICAL TRIAL: NCT04668261
Title: Longitudinal Investigation of Brain Blood Flow Changes in Neurosurgical Patients
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02314
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Brain Blood Flow Impairment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurosurgical patients: • Neurosurgical diseases with the potential to alter blood flow to the brain:
  * Cerebrovascular disease
  * Brain tumors
  * Normal Pressure Hydrocephalus
  Interventions: Other: Advanced imaging investigation
- Healthy subjects: * Male and Female subjects >18 years of age
  * Written Informed Consent by the participant after information about the project. Foreign speaking healthy subjects should be accompanied by a person with sufficient German language proficiency to act as a translator
  Interventions: Other: Advanced imaging investigation

INTERVENTIONS:
Other: Advanced imaging investigation — MRI imaging

SUMMARY:
Primary study objective:

• Longitudinal observation of brain blood flow changes in neurosurgical patients with or without a neurosurgical intervention as compared to a healthy cohort.

Secondary study objectives:

* Longitudinal observation of hemodynamic patterns versus structural brain tissue changes in neurosurgical patients.
* Changes in blood flow patterns and structural brain tissue after neurosurgical interventions as compared to a healthy cohort.
* Determining hemodynamic imaging patterns that can be tested as novel imaging markers.

DETAILED DESCRIPTION:
Primary study objective:

• to study the longitudinal observation of brain blood flow changes in neurosurgical patients to evaluate the effect of surgical or conservative treatment on the brain structural and hemodynamic integrity.

Secondary study objectives:

* To observe the relationship between longitudinal changes in hemodynamic patterns and structural brain tissue changes in neurosurgical patients.
* To determine different hemodynamic patterns that may be used as novel imaging biomarkers in future studies.

4.2 Outcomes

Outcomes of the project:

Primary endpoint:

To find correlation between course of disease, neurosurgical intervention and changes in brain blood flow and brain structure.

Secondary endpoints:

* Correlation between progression of disease and hemodynamic patterns over time (ie. novel imaging markers)
* Correlation of clinical management (neurosurgical treatment vs. best medical care) and changes in brain blood flow.

ELIGIBILITY:
Inclusion criteria

Patients:

* Male and Female subjects >18 years of age
* Written informed consent after participants' information. Foreign speaking patients should be accompanied by a person with sufficient German language proficiency to act as a translator
* Neurosurgical diseases with the potential to alter blood flow to the brain:

  * Cerebrovascular disease
  * Brain tumors
  * Normal Pressure Hydrocephalus

Healthy subjects:

* Male and Female subjects >18 years of age
* Written Informed Consent by the participant after information about the project. Foreign speaking healthy subjects should be accompanied by a person with sufficient German language proficiency to act as a translator

Exclusion criteria:

Patients:

* Unwilling or unable to co-operate with breathing maneuvers
* Respiratory or cardiac limitations to breathing through a mask
* Medical contra-indications to limited hypercapnia (high CO2 - 50 mmHg) or hypocapnia (low CO2 - 30 mmHg) (i.e., known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Standard contraindications for MRI scanning
* Verbal confirmed pregnancy
* Known multiple intracranial diseases
* Presence of intracranial hemorrhage within the last 3 months
* Symptomatic increased intracranial pressure

Healthy subjects:

* Unwilling or unable to co-operate with breathing maneuvers
* Respiratory or cardiac limitations to breathing through a mask
* Medical contra-indications to limited hypercapnia (high CO2 - 50 mmHg) or hypocapnia (low CO2 - 30 mmHg) (i.e., known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Standard contraindications for MRI scanning
* Verbal confirmed pregnancy
* Anamnesticly a history of neurological disease or current neurological deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurosurgical patients with the potential to have altered blood flow to the brain
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
• Longitudinal observation of brain blood flow changes in neurosurgical patients with or without a neurosurgical intervention as compared to a healthy cohort. | 5 years
  blood flow changes will be assessed with quantitative blood oxygenation-level dependent cerebrovascular reactivity measurements

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided